CLINICAL TRIAL: NCT03187990
Title: Single-center Study for Biopsy Guidance Using Gallium-68 Labeled Prostate-specific Membrane Antigen (PSMA) PET/MRI in Patients With Elevated PSA Eligible for Prostate Biopsy in Comparison to Multiparametric MRI.
Brief Title: Positron Emission Tomography / Magnetic Resonance Imaging (PET/MRI) Guided Biopsy in Men With Elevated PSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Irene Burger (Other)
Responsible Party: Sponsor-Investigator, Irene Burger, Principal investigator, University of Zurich
Organization: University of Zurich (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KEK-ZH-NR: 2017-00016
Record Dates: First submitted 2017-06-13; First posted 2017-06-15 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-08

CONDITIONS: Prostate Cancer
Keywords: PSMA PET/MRI; Guided Biopsy; Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — gallium 68 PSMA-11

STUDY DESIGN:
Intervention Model Description: In both arms PET/MR is compared to mpMRI for diagnostic accuracy for PCA detection.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PET/MRI before biopsy (Experimental): Patients with suspected areas on mpMRI will undergo additional [68Ga]PSMA-11 PET/MRI scan with subsequent mpMRI and PET/MRI guided biopsy.
  Interventions: Drug: [68Ga]PSMA-11; Drug: [18F]PSMA-1007
- PET/MRI after biopsy (Experimental): Patients with unclear areas or a negative finding in the mpMRI for MRI guided biopsy but positive biopsy, which will undergo the additional [68Ga]PSMA-11 PET/MRI scan with [68Ga]PSMA.
  Interventions: Drug: [68Ga]PSMA-11

INTERVENTIONS:
Drug: [68Ga]PSMA-11 — PET/MRI with [68Ga]PSMA will be compared to mpMRI for biopsy guidance.
  Other Names: PSMA PET/MRI
Drug: [18F]PSMA-1007 — 18F-PSMA-1007 PET/CT for biopsy guidance and intraoperative target verification.
  Other Names: PSMA PET/CT
  Arms: PET/MRI before biopsy

SUMMARY:
In 22% of patients with elevated Prostate-specific antigen (PSA) MRI guided biopsy will not detect significant prostate cancer (PCA) (defined as either: Gleason score (GS) ≥ 3+4 or tertiary pattern 5, or final stage ≥ pT3a and/or pN1). Therefore this study evaluates the ability of [68Ga]PSMA PET/MRI to detect and localize significant primary PCA to accurately direct prostate needle biopsy using the Gleason score from the histology of the core biopsies as standard of truth.

DETAILED DESCRIPTION:
In this open label, single center, non-randomized, diagnostic study we plan to include 40 men with elevated PSA (ages 30-50 PSA >2.5 ng/mL; ages 50-80 PSA > 4ng/mL), which are assigned to a MRI guided biopsy.

These patients will undergo one additional PET/MRI scan with [68Ga]PSMA within two to three weeks before the biopsy (Arm A), or in case of an unclear/negative MRI scan but positive biopsy two to three weeks after biopsy (Arm B). In Arm A a radiologist will delineate the suspected areas on (A) multiparametric magnetic resonance image (mpMRI) and a nuclear medicine physician will delineate and color code the suspicious areas on the PET/MRI: (B) [68Ga]PSMA. The images will be loaded into the BiopSee® system. Lesions positive on both modalities will be labeled as "AB". Every suspicious lesion will be targeted with 3 cores. A maximum of 3 targets will be selected per patient.

For arm B: PET/MRI results will be correlated with the template biopsy results.

The data analysis of Arm A and Arm B will be identical. For the analysis the Gleason score from the histology of the core biopsies will serve as standard of truth.

After completion of the PET/MR study part - an amendment for PET/CT was submitted to the local ethics commity and acknowledged to include 10 more participants with PSMA PET/CT to investigate the use of PET/CT guided biopsy and intraoperative verivication of the target with a gamma counter.

ELIGIBILITY:
Inclusion Criteria:

1. Previously undiagnosed patients with elevated PSA (ages 30-50 PSA >2.5 ng/mL; ages 50-80 PSA > 4ng/mL), eligible for prostate needle biopsy.
2. Patients can have negative prior needle biopsy(ies) for suspected prostate cancer
3. mpMRI with at least one suspicious target lesion (Arm A), or negative mpMRI but positive biopsy (Arm B).
4. Written informed consent
5. Age > 30

Exclusion Criteria:

1. Age> 80
2. Contraindication to MRI or prostate biopsy (e.g. extreme claustrophobia, metallic implants incompatible with MRI, anatomical contraindications, coagulopathy, severe medical comorbidity prohibiting halting of anticoagulation therapies)
3. Active urinary tract infection or indwelling catheter
4. Prior pelvic irradiation
5. Prior prostatectomy
6. Prior androgen deprivation hormonal therapy
7. Prostate biopsy within 8 weeks prior to study
8. Prior transurethral resection of the prostate (TURP)

Ages: 30 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2017-03-03 (Actual); Primary Completion 2021-08-03 (Actual); Study Completion 2021-08-03 (Actual)

PRIMARY OUTCOMES:
Rate of positive histopathology for [68Ga]PSMA-11 positive lesions | 7 months
  PCA detection of PET/MRI versus mpMRI based on histopathology per patient and per prostate section.

SECONDARY OUTCOMES:
Correlation of [68Ga]PSMA-11 with tumor aggressiveness | 7 months
  Correlation of stanadized uptake value (SUV) on [68Ga]PSMA-11 with Gleason Score on histopathology.

CONTACTS AND LOCATIONS:
Overall Officials: Irene A Burger, MD, Principal Investigator — UniversitaetsSpital Zuerich
Locations (1):
- University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ferraro DA, Laudicella R, Zeimpekis K, Mebert I, Muller J, Maurer A, Grunig H, Donati O, Sapienza MT, Rueschoff JH, Rupp N, Eberli D, Burger IA. Hot needles can confirm accurate lesion sampling intraoperatively using [18F]PSMA-1007 PET/CT-guided biopsy in patients with suspected prostate cancer. Eur J Nucl Med Mol Imaging. 2022 Apr;49(5):1721-1730. doi: 10.1007/s00259-021-05599-3. Epub 2021 Nov 2. PMID 34725726
- [Derived] Ferraro DA, Becker AS, Kranzbuhler B, Mebert I, Baltensperger A, Zeimpekis KG, Grunig H, Messerli M, Rupp NJ, Rueschoff JH, Mortezavi A, Donati OF, Sapienza MT, Eberli D, Burger IA. Diagnostic performance of 68Ga-PSMA-11 PET/MRI-guided biopsy in patients with suspected prostate cancer: a prospective single-center study. Eur J Nucl Med Mol Imaging. 2021 Sep;48(10):3315-3324. doi: 10.1007/s00259-021-05261-y. Epub 2021 Feb 23. PMID 33620559